CLINICAL TRIAL: NCT05094622
Title: Physical Exercise in Patients With Postural Orthostatic Tachycardia Syndrome (POTS) After Covid-19.
Brief Title: Physical Training in Patients With POTS After Covid-19
Acronym: POTS-ReCOV
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Collaborators: Karolinska University Hospital (Other)
Responsible Party: Principal Investigator, Malin Nygren-Bonnier, Physiotherapist, Senior lecturer and Associate Professor, Karolinska Institutet
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: POTS-ReCov
Record Dates: First submitted 2021-10-25; First posted 2021-10-26 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-04

CONDITIONS: Covid19; Post-acute Covid-19 Syndrome; Postural Orthostatic Tachycardia Syndrome
Keywords: physiotherapy; rehabilitation; physical exercise; quality of life; physical activity
MeSH Terms: conditions — COVID-19; Post-Acute COVID-19 Syndrome; Postural Orthostatic Tachycardia Syndrome; Motor Activity

STUDY DESIGN:
Intervention Model Description: single subject design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Physical exercise (Experimental): Physical exercise program
  Interventions: Other: Physical exercise program

INTERVENTIONS:
Other: Physical exercise program — A specially designed exercise training program based on a previous study. The intervention of physical exercise will consist of different exercises to enhance muscle strength and endurance and will be individually adjusted and start in a different position with a progression in dose, intensity, and position. It will be performed 3 times /week during a period of 12-20 weeks.

SUMMARY:
Covid-19 has the potential to affect physical, cognitive and psychological functions in multiple ways. It has been clear that a significant proportion of patients with Covid-19 develop long-term symptoms. The term post-acute Covid-19 syndrome (PACS) is now used to describe the wide range of prolonged symptoms following the infection. Patients may need specialized rehabilitation to be able to meet the complex symptoms and problems that may arise. A more specific syndrome that seems to occur more frequently than expected in the group of non-hospitalized patients who have had Covid-19 is the postural orthostatic tachycardia syndrome (POTS).

To evaluate the effects of physical training in patients with POTS after Covid-19 a single subject design will be used (the patient is their own control). Inidividual semistructured interviews will be performed to explore and describe the patients´ experiences of the rehabilitation intervention.

Participants: Patients diagnosed with POTS after Covid-19 (N=30) will be included.

Procedure and outcomes: The primary outcomes are physical activity and health-related quality of life. Secondary outcomes are: physical capacity, active standing test, Malmö-POTS-questionnaire, Anxiety and depression, fatigue, self-reported outcome measure of physical function and work ability.

Initially measurements will be performed several times during a period of 2-4 weeks to obtain a baseline before the intervention starts. Then the included participants will undergo a specially designed physical training program that will be performed 3 times /week during a period of 12 weeks. The intervention of physical training will consist of different exercises to enhance muscle strength and endurance. The intervention will be individually adjusted with a progression in dose, intensity, and position. The exercise is based on a program used in a previous study. Measurements will then be repeated after completion of the intervention period.

A qualitative approach, with semistructured interviews, will be used to explore the patients´ experiences of the intervention, after commence of the interventional trial.

DETAILED DESCRIPTION:
Introduction:

Covid-19 was declared a global pandemic in March 2020 by the World Health Organization (WHO). In August 2021, in Sweden, over 1 100 000 cases were confirmed and over 14 000 deaths. Initially, it was suspected that Covid-19 would primarily affect the airways, but several studies have now shown that it is a disease with multisystem manifestations. The impact of the virus ranges from an asymptomatic infection to a severe and life-threatening disease that can affect the cardiac, renal gastrointestinal, nervous, endocrine, and musculoskeletal systems. Therefore, Covid-19 has the potential to affect physical, cognitive, and psychological functions in multiple ways. It has been clear that a significant proportion of patients with Covid-19 develop long-term symptoms. Signs and symptoms may arise from any system in the body, often with significant overlap, and may develop over time. The term post- acute Covid-19 syndrome (PACS) is now used to describe the wide range of prolonged symptoms following the infection.

Fatigue, decreased physical and psychological function have been reported in the initial recovery phase, but still little is known on the long-term consequences. Patients who have been in hospital for Covid-19 for a long time may need specialized rehabilitation, however, also non-hospitalized patients with mild symptoms may need specific rehabilitation to be able to meet the complex symptoms and problems that may arise. Previous studies on the recovery and rehabilitation after other coronavirus shows the importance to develop tailored interventions so that these patients receive appropriate rehabilitation with a multi-professional approach throughout the whole care chain. Some studies suggest that the rehabilitation should be similar to pulmonary rehabilitation, but since a lot of patients often have symptoms from different organ systems this is not yet fully investigated and needs to be addressed from different perspectives.

A more specific syndrome that seems to occur more frequently than expected in persons who have had Covid-19 is the postural orthostatic tachycardia syndrome (POTS). It is a form of chronic orthostatic intolerance in which upright posture is associated with an excessive increase in heart rate (HR) with a >6-month history of symptoms. Patients with POTS may have problems associated to the diagnoses, such as palpitation exercise intolerance, hypermobile joints, exercise intolerance, migraine headaches, brain-fog, sleep disturbances, and fatigue. Symptoms that can be exacerbated by simple activities of daily life and exercise. Consequently, patients seem to reduce their physical activity, which might reduce their physical capacity and function and thus limit activities in daily living.

Nevertheless, supervised individual tailored physical exercises, is a recommended non-pharmacological treatment of POTS. However, few studies have investigated the effect of physical exercise in POTS, and to date, no studies have evaluated the effect of individually tailored rehabilitation in persons with POTS after Covid-19.

At the Karolinska University Hospital there is a specialized multidisciplinary and multi-professional approach aiming to follow up hospitalized patients and non-hospitalized persons (referrals from primary care) with PACS.

This study is part of a bigger research project (ReCOV) and is integrated with the clinical follow-up and linked research project of patients who have been hospitalized or reffered to the clinic from primary care.

The hypothesis is that a individually tailored rehabilitation program will have an effect on HRQoL and physical activity for individuals with POTS after Covid-19.

The overall aim of this study is to evaluate the effects of an individually tailored rehabilitation program and its impact on health-related quality of life (HRQoL), physical activity, physical and psychological function and work ability in persons with POTS after Covid-19. Furthermore, to explore and describe the patients´ experiences of the rehabilitation intervention.

Methods:

A) To evaluate the effects of physical training in patients with POTS after Covid-19 a single subject design will be used (the patient is their own control).

B) A qualitative approach with inidividual semistructured interviews will be performed with a strategic sample of patients´ to explore their experiences of the rehabiliation intervention.

Participants:

A) A total of 30 patients, diagnosed with POTS after Covid-19, will be recruited at the outpatient clinic at Karolinska University Hospital.

B) A strategic sample will be applied with the aim of selecting persons representing varied characteristics regarding gender, age, professions, level of disability and living conditions

Procedure and outcomes:

A) The primary outcomes are physical activity (ActivPal accelerometer) and health-related quality of life (EQ-5D-5L). The secondary outcomes are 6 minute walk test, physiological responses during an active standing test, Malmö-POTS-questionnaire, anxiety and depression questionnaires (GAD-7 and PHQ-9), fatigue questionnaire (FSS), self-reported outcome measure of physical function (PSFS) and the work ability (WAI) questionnaire.

Initially measurements will be performed several times during a period of 2-4 weeks to obtain a baseline before the intervention starts. Thereafter, the included participant will undergo a specially designed physical training program that will be performed 3 times /week during a period of 12 weeks and will take place at the physiotherapy outpatient clinic at the hospital, or at primary care facility or at home. The intervention of physical training will consist of different exercises to enhance muscle strength and endurance. The intervention will be individually adjusted and tailored (by a physiotherapist) with a progression in dose, intensity and position. The exercise is based on a program used in a previous study (se references below). Measurements will then be repeated, during a period of 1-2 weeks, after completion of the intervention period.

Demographic data and data on feasibility (acceptance of the program, adverse events etc) and outcome variables will be collected.

B). Semi-structured interviews will be conducted after commencing of the intervention. An interview-guide with open-ended and probing questions focusing on participants´ experiences of participating in the intervention and the impact on their everyday life and physical activity. All interviews will be audio-recorded, and then transcribed by a professional transcriber. The interviews are estimated to take 30 to 60 minute and the participants can choose whether they want to be interviewed by phone, digital meeting, or a physical meeting.

Data analyses:

A). This is a multiple single case study with A-B-design. This will allow for analyses with randomization testing and meta-analytical approaches to evaluate the effect of the intervention. With several measuring points and 30 participant the investigators estimate to have sufficient power in relation to design and analyses plan and research questions. Data will be described with mean (standard deviation), median (inter-quartile range) and proportion and analyzed with parametric and non-parametric methods depending on data level and analysis will be performed to compare differences between the baseline data and data from the intervention-period.

B). The interviews will be verbatim transcribed (in their entirety) and analyzed through an inducive content analysis, an appropriate method for identifying, organizing, and categorizing the content of a narrative text in a systematic way.

Clinical significance:

Covid-19 is a new disease and large knowledgegaps need to be filled. The orthostatic intolerance, migraine, palpitations, fatigue and other symptoms connected to POTS after Covid-19, has the potential to affect physical, cognitive, and psychological functions in multiple ways and lead to longer periods of sick-leave, and a negative impact on health related quality of life in the long-term perspective. Therefore, development of a rehabilitation program with specific tailored interventions will be necessary to improve physical and psychological function, as well as health-related quality of life and work ability.

Few studies have investigated the effect of physical exercise in POTS, and to date, no studies have evaluated the effect of physical exercise following covid-19 infection in POTS. There is an urgent need to develop individual rehabilitation interventions, targeting these symptoms. Moreover, to increase knowledge about how individualized rehabilitation interventions leads to physical and mental improvements improvements in patients, It is of great importance that data is collected systematically and standardized. If significant effects occur, the possibility to generalize the results to other individuals with Covid-19, are promising. The physical interventions may thus improve the ability to adjust to the implications of Covid-19, which can potentially have significant health economic effects. For example, the interventions may prolong patients' meaningful activities of daily living and their ability to return to their previous workplaces (conduct their professions). This project will deepen the knowledge about the effects of specialized rehabilitation. The new knowledge generated by this project will be of great benefit to the large number of patients affected by this new global disease.

Ethical considerations:

The project has been approved by the Swedish Ethical Review Authority. The participants will receive verbal and written information about the study and informed consent will be obtained from all participants.

ELIGIBILITY:
Inclusion Criteria: Adult patients (>18 years) diagnosed with postural orthostatic tachycardia syndrome after Covid-19.

Exclusion Criteria: Patient not able to perform the intervention due to cognitive or physical dysfunction, Already on-going physical intervention.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-01-10 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Change in Health-Related Quality of Life (HRQoL) | Measured before and after the intervention period of 12-16 weeks to detect a change
  Measured with EuroQualityOf Life 5 dimensions questionnaire (EQ-5D-5L), which is an instrument that evaluates the generic quality of life. EQ-5D includes a descriptive system, which comprises 5 dimensions of health: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. A descriptive index-score between 0-1, higher score indicates higher HRQoL. EQ-5D also includes a visual analog scale (VAS), which records the respondent's self-rated health status on a graduated (0-100) scale, with higher scores for higher HRQoL.
Change in time in upright position and steps per day | Measured before and after the intervention period of 12-16 weeks to detect a change
  Measured with two accelerometers attached to upper and lower limbs to measure time (hours, minutes) in upright position during 7 consecutive days

SECONDARY OUTCOMES:
Change in walking distance during 6 minute walk test | Measured before and after the intervention period of 12-16 weeks to detect a change
  Change in walking distance measured in meters during 6 minutes walk test (6MWT)
Change in oxygen saturation during 6 minute walk test | Measured before and after the intervention period of 12-16 weeks to detect a change
  Change in the lowest oxygen saturation level measured in percentage (%) with pulse oximetry during 6 minute walk test.
Change in oxygen desaturation during 6 minute walk test | Measured before and after the intervention period of 12-16 weeks to detect a change
  Change in drop in percentage points in oxygen saturation during 6 minute walk test. The drop in percentage points is calculated by subtracting the oxygen level at rest before the test with the lowest level during the test.
Change in dyspnea during 6 minute walk test | Measured before and after the intervention period of 12-16 weeks to detect a change
  Change in perceived dyspnea measured with Borg Category-Ratio scale (Borg CR-10) at the end of 6 minute walk test. Borg CR-10 ranging between 0-10. The higher the score, the higher the dyspnea.
Change in leg fatigue during 6 minute walk test | Measured before and after the intervention period of 12-16 weeks to detect a change
  Change in perceived leg fatigue measured with Borg CR-10 at the end of 6 minute walk test. Borg CR-10 ranging between 0-10. The higher the score, the higher the leg fatigue.
Change in exertion during 6 minute walk test | Measured before and after the intervention period of 12-16 weeks to detect a change
  Change in perceived exertion measured with Borg Rating of Perceived Exertion (Borg RPE) at the end of 6 minutes walk test. Borg RPE ranging between 6-20. The higher the score, the higher the exertion.
Change in heart rate during 6 minute walk test | Measured before and after the intervention period of 12-16weeks to detect a change
  Change in the highest heart rate measured in beats per minute with pulse oximeter during 6 minute walk test
Change in Self-reported POTS-symptoms | Measured before and after the intervention period of 20 weeks to detect a change
  Measured with Malmö-POTS-questionnaire (MaPS), which is a self assessment tool examining common symptoms in POTS. MaPS consists of 12 items. Patients are asked to rate symptoms on a scale from 0-10 on each item. 0 i= no symptom and 10 = worst imaginable. Total score ranging from 0-120. Higher score indicates more POTS-symptoms.
Change in Anxiety - Generalised Anxiety Disorder 7-item scale | Measured before and after the intervention period of 12-16 weeks to detect a change
  Measured with Generalised Anxiety Disorder 7-item scale (GAD-7) which is a self assessment tool. Total score ranging from 0-21. Higher score indicates higher anxiety.
Change in Depression - Patient Health Questionnaire-9 | Measured before and after the intervention period of 12-16 weeks to detect a change
  Measured with Patient Health Questionnaire-9 (PHQ-9). PHQ-9 which contains 9 items. Total score ranges from 0 to 27. Higher score indicate more severe depression symptoms.
Change in Fatigue | Measured before and after the intervention period of 12-16 weeks to detect a change
  Measured with Fatigue Severity Scale (FSS), which is a 9-item scale that measures the severity of fatigue and its effect on a person's activities and lifestyle in patients with a variety of disorders. Total score ranging from 9-63. The higher the score, the more severe the fatigue is.
Change in Work ability | Measured before and after the intervention period of 12-16 weeks to detect a change
  Measured with percentage of full-time work ability and Work Ability Index (WAI). WAI is a self assessment tool consisting of 7 items. Scores ranging from 7-49. Higher score indicates higher work ability.
Change in Self-reported outcome measure of physical function | Measured before and after the intervention period of 12-16 weeks to detect a change
  Measured with Patient Specific Functional Scale (PSFS), a questionnaire that can be used to quantify activity limitation and measure functional outcome for patients. Patients are asked to identify three to five important activities they are unable to perform or are having difficulty with because of their problem. In addition to identifying the activities, patients are asked to rate, on a scale ranging from 0-10, the current level of difficulty associated with each activity. The higher the score, the less difficulty to perform the activity.
Change in blood pressure during Active standing test | Measured before and after the intervention period of 12-16 weeks to detect a change
  Measured with Active standing test according to a specific protocol with measurements of responses in systolic and diastolic blood pressure after getting up to standing from the supine position.
Change in heart rate response during Active standing test | Measured before and after the intervention period of 12-16 weeks to detect a change
  Measured with Active standing test according to a specific protocol with measurements of responses in heart rate after getting up to standing from the supine position.
Change in oxygen saturation during Active standing test | Measured before and after the intervention period of 12-16 weeks to detect a change
  Measured with Active standing test according to a specific protocol with measurements of responses in oxygen saturation, measured with pulse oximetry, after getting up to standing from the supine position.
Change in dyspnea during Active standing test | Measured before and after the intervention period of 12-16 weeks to detect a change
  Measured with Active standing test according to a specific protocol with measurements of responses in perceived dyspnea measured with Borg CR-10 scale after getting up to standing from the supine position.
Change in exertion during Active standing test | Measured before and after the intervention period of 12-16 weeks to detect a change
  Measured with Active standing test according to a specific protocol with measurements of responses in perceived exertion with Borg RPE scale after getting up to standing from the supine position.
Change in Physical activity | Measured before and after the intervention period of 12-16 weeks to detect a change
  Measured with Frändin/Grimby activity scale, which is a self-assessment scale about current levels of physical activity, ranging from 1 to 6. The higher the score, the higher the level of physical activity.
Change in orthostatic symptoms | Measured before and after the intervention period of 12-16 weekt to detect a change
  Assessed with the Vanderbilt Orthostatic Symptom Scale (VOSS). After the Active standing test (AST) the participant uses a self-assessment questionnaire about orthostatic symptoms prominent during the Active standing test (performed according to a specific protocol with measurements of responses in systolic and diastolic blood pressure after getting up to standing from the supine position). The scale range from 0=no symptoms, to 10=worst imaginable symptoms. The scale includes 9 items regarding orthostatic symptoms and the higher the score, the higher level of symptoms during the orthostatic test.

CONTACTS AND LOCATIONS:
Overall Officials: Malin Nygren Bonnier, PhD, Principal Investigator — Karolinska Institutet
Locations (1):
- Karolinska University Hospital, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fu Q, Levine BD. Exercise and non-pharmacological treatment of POTS. Auton Neurosci. 2018 Dec;215:20-27. doi: 10.1016/j.autneu.2018.07.001. Epub 2018 Jul 4. PMID 30001836
- [Background] Crook H, Raza S, Nowell J, Young M, Edison P. Long covid-mechanisms, risk factors, and management. BMJ. 2021 Jul 26;374:n1648. doi: 10.1136/bmj.n1648. PMID 34312178
- [Background] Nalbandian A, Sehgal K, Gupta A, Madhavan MV, McGroder C, Stevens JS, Cook JR, Nordvig AS, Shalev D, Sehrawat TS, Ahluwalia N, Bikdeli B, Dietz D, Der-Nigoghossian C, Liyanage-Don N, Rosner GF, Bernstein EJ, Mohan S, Beckley AA, Seres DS, Choueiri TK, Uriel N, Ausiello JC, Accili D, Freedberg DE, Baldwin M, Schwartz A, Brodie D, Garcia CK, Elkind MSV, Connors JM, Bilezikian JP, Landry DW, Wan EY. Post-acute COVID-19 syndrome. Nat Med. 2021 Apr;27(4):601-615. doi: 10.1038/s41591-021-01283-z. Epub 2021 Mar 22. PMID 33753937
- [Background] Fedorowski A. Postural orthostatic tachycardia syndrome: clinical presentation, aetiology and management. J Intern Med. 2019 Apr;285(4):352-366. doi: 10.1111/joim.12852. Epub 2018 Nov 23. PMID 30372565
- [Background] Johansson M, Stahlberg M, Runold M, Nygren-Bonnier M, Nilsson J, Olshansky B, Bruchfeld J, Fedorowski A. Long-Haul Post-COVID-19 Symptoms Presenting as a Variant of Postural Orthostatic Tachycardia Syndrome: The Swedish Experience. JACC Case Rep. 2021 Apr;3(4):573-580. doi: 10.1016/j.jaccas.2021.01.009. Epub 2021 Mar 10. PMID 33723532
- [Background] Stahlberg M, Reistam U, Fedorowski A, Villacorta H, Horiuchi Y, Bax J, Pitt B, Matskeplishvili S, Luscher TF, Weichert I, Thani KB, Maisel A. Post-COVID-19 Tachycardia Syndrome: A Distinct Phenotype of Post-Acute COVID-19 Syndrome. Am J Med. 2021 Dec;134(12):1451-1456. doi: 10.1016/j.amjmed.2021.07.004. Epub 2021 Aug 11. PMID 34390682
- [Background] Arnold AC, Ng J, Raj SR. Postural tachycardia syndrome - Diagnosis, physiology, and prognosis. Auton Neurosci. 2018 Dec;215:3-11. doi: 10.1016/j.autneu.2018.02.005. Epub 2018 Feb 28. PMID 29523389
- [Background] Benrud-Larson LM, Dewar MS, Sandroni P, Rummans TA, Haythornthwaite JA, Low PA. Quality of life in patients with postural tachycardia syndrome. Mayo Clin Proc. 2002 Jun;77(6):531-7. doi: 10.4065/77.6.531. PMID 12059122